CLINICAL TRIAL: NCT01812551
Title: Osteoporosis in Cystic Fibrosis: Study of Bone Mass and Bone Metabolism, and Prospective Randomized Therapeutic Trial.
Brief Title: Treatment of Low Bone Density in Cystic Fibrosis.
Acronym: OSCYF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Fondazione Telethon (Other)
Responsible Party: Principal Investigator, Maria Luisa Bianchi, MD, First level manager, Istituto Auxologico Italiano
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02A001
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Osteoporosis; Cystic Fibrosis
Keywords: cystic fibrosis; children; adolescents; low bone mass; osteoporosis; alendronate; fractures
MeSH Terms: conditions — Osteoporosis; Cystic Fibrosis; Fractures, Bone | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alendronate (Active Comparator): 128 subjects participated in the study's Phase 2 (1-year double-blind, randomized, placebo-controlled, parallel group study).
  65 subjects were randomized to this arm. Oral alendronate dose: 5 mg/day, if body weight ≤25 kg; 10 mg/day, if body weight >25 kg.
  Interventions: Drug: Alendronate
- Placebo (Placebo Comparator): 128 subjects participated in the study's Phase 2 (1-year double-blind, randomized, placebo-controlled, parallel group study).
  63 subjects were randomized to this arm. Oral placebo (inactive pills).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alendronate — As active drug, we used Alendros (Abiogen Pharma, Pisa, Italy), distributed to the patients in plain bottles and boxes (bearing only the center and patient codes).
  Other Names: Alendros
  Arms: Alendronate
Drug: Placebo — Placebo was distributed to the patients in plain bottles and boxes (bearing only the center and patient codes).
  Arms: Placebo

SUMMARY:
Cystic fibrosis (CF) -- an autosomal recessive genetic disease affecting about 60,000 individuals worldwide, including about 3,800 in Italy -- is often associated with low bone mineral mass. The current aggressive therapies have ensured a much longer survival of CF patients but this has led to a higher frequency of osteoporosis and bone fractures, a serious problem which not only affects quality of life, but also hinders further therapeutic measures.

The aim of this study, conducted on a large group of children, adolescents and young adults with CF, has been the evaluation of bone mass changes after 1 year of a simple treatment with RDA-adjusted dietary calcium plus 25-OH vitamin D supplementation, and the feasibility and efficacy of alendronate treatment (for another year) in patients not responding to calcium + 25-OH vitamin D alone.

DETAILED DESCRIPTION:
The study included 2 phases.

Phase 1 (1-year open-label observational study): following baseline evaluation, bone mass changes have been studied with a simple therapy of adequate calcium intake and 25-OH vitamin D supplements in all eligible subjects (N=171).

Phase 2 (1-year double-blind, randomized, placebo-controlled, parallel group study): the 128 subjects showing an insufficient response to calcium + 25-OH vitamin D alone (bone mass increase <5%) at the end of Phase 1, were randomized into 2 groups and assigned to alendronate treatment (N=65) or placebo (N=63) (in addition to calcium and 25-OH vitamin D as during Phase 1).

The study has been carried out by the Coordinator's Institution (Istituto Auxologico Italiano)in collaboration with most Regional Reference Centers for CF in Italy.

ELIGIBILITY:
Inclusion Criteria:

* age 2-30 years
* clinically stable condition
* regular menses in females
* low Bone Mineral Apparent Density for age (defined as BMAD Z-score ≤-2.0 if age ≤18 years or ≤-2.5 if age >18 years).

Exclusion Criteria:

* two or more episodes of hypercalcemia and/or hypercalciuria
* contraindications to 25-OH vitamin D or alendronate treatment
* recent transplantation
* other diseases or medications (glucocorticoids excepted) associated with bone loss.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 171 (Actual)
Dates: Start 2002-10; Primary Completion 2006-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral density increase at lumbar spine. | up to 24 months
  Bone mineral density evaluated by DXA. Bone mineral apparent density calculated to correct for bone size (growing subjects). Z-score calculated.
  Measurements: Phase 1 (171 subjects): Baseline, 6 months, 12 months. Phase 2 (128 subjects, randomized to 2 arms: placebo or alendronate): 18 months, 24 months.

SECONDARY OUTCOMES:
Changes in bone turnover markers. | baseline and up to 24 months
  Bone turnover markers: (serum) osteocalcin (OC), bone specific alkaline phosphatase (BSAP), C-terminal telopeptide of procollagen 1 (CTx); (urine) terminal telopeptide of procollagen 1 (NTx).
Fracture rate. | at 12th and 24th month
  Appendicular fractures were evaluated at baseline (previous fractures) and throughout the 2 years of study (incident fractures) with X-rays.
  Vertebral fractures were evaluated at the end of Phase 1 (12th month) and at the end of Phase 2 (24th month) with lateral thoracic and lumbar spine X-rays.
Adverse effects of alendronate. | continuously throughout Phase 2 (2nd year of study)
  Evaluated on the basis of lab tests (calcemia, calciuria, blood cell count, liver and kidney function), FEV1 changes, and other signs/symptoms (e.g. pain, fever, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Bianchi, M.D., Principal Investigator — Istituto Auxologico Italiano
Locations (11):
- CRR Fibrosi Cistica, Divisione Gastroenterologia, Ospedale Bambin Gesù, Vatican City, Holy See
- Italy (10):
  - CRR Fibrosi Cistica, Unità Operativa di Pediatria, Ospedale Misericordia, Grosseto
  - CRR Fibrosi Cistica, Clinica Pediatrica, Policlinico Universitario di Messina, Messina
  - Istituto Auxologico Italiano IRCCS, Milan
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Università degli Studi di Milano, Milan
  - CRR Fibrosi Cistica, Dipartimento Pediatria, Università Federico II, Napoli
  - CRR Fibrosi Cistica Adulti, Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano
  - CRR Fibrosi Cistica, Ospedale dei Bambini, ARNAS Civico, Palermo
  - CRR Fibrosi Cistica, Dipartimento di Pediatria, Policlinico Umberto I, Roma
  - CRR Fibrosi Cistica, Divisione di Pediatria, Istituto Burlo Garofolo, Trieste
  - CRR Fibrosi Cistica, Azienda Ospedalierouniversitaria di Verona, Verona

REFERENCES:
- [Background] Grey AB, Ames RW, Matthews RD, Reid IR. Bone mineral density and body composition in adult patients with cystic fibrosis. Thorax. 1993 Jun;48(6):589-93. doi: 10.1136/thx.48.6.589. PMID 8346485
- [Background] Henderson RC, Madsen CD. Bone density in children and adolescents with cystic fibrosis. J Pediatr. 1996 Jan;128(1):28-34. doi: 10.1016/s0022-3476(96)70424-9. PMID 8551418
- [Background] Bhudhikanok GS, Lim J, Marcus R, Harkins A, Moss RB, Bachrach LK. Correlates of osteopenia in patients with cystic fibrosis. Pediatrics. 1996 Jan;97(1):103-11. PMID 8545201
- [Background] Baroncelli GI, De Luca F, Magazzu G, Arrigo T, Sferlazzas C, Catena C, Bertelloni S, Saggese G. Bone demineralization in cystic fibrosis: evidence of imbalance between bone formation and degradation. Pediatr Res. 1997 Mar;41(3):397-403. doi: 10.1203/00006450-199703000-00016. PMID 9078542
- [Background] Humphries IR, Allen JR, Waters DL, Howman-Giles R, Gaskin KJ. Volumetric bone mineral density in children with cystic fibrosis. Appl Radiat Isot. 1998 May-Jun;49(5-6):593-5. doi: 10.1016/s0969-8043(97)00203-0. No abstract available. PMID 9569551
- [Background] Aris RM, Renner JB, Winders AD, Buell HE, Riggs DB, Lester GE, Ontjes DA. Increased rate of fractures and severe kyphosis: sequelae of living into adulthood with cystic fibrosis. Ann Intern Med. 1998 Feb 1;128(3):186-93. doi: 10.7326/0003-4819-128-3-199802010-00004. PMID 9454526
- [Background] Bhudhikanok GS, Wang MC, Marcus R, Harkins A, Moss RB, Bachrach LK. Bone acquisition and loss in children and adults with cystic fibrosis: a longitudinal study. J Pediatr. 1998 Jul;133(1):18-27. doi: 10.1016/s0022-3476(98)70172-6. PMID 9672505
- [Background] Henderson RC, Madsen CD. Bone mineral content and body composition in children and young adults with cystic fibrosis. Pediatr Pulmonol. 1999 Feb;27(2):80-4. doi: 10.1002/(sici)1099-0496(199902)27:23.0.co;2-j. PMID 10088930
- [Background] Bianchi ML, Cimaz R, Bardare M, Zulian F, Lepore L, Boncompagni A, Galbiati E, Corona F, Luisetto G, Giuntini D, Picco P, Brandi ML, Falcini F. Efficacy and safety of alendronate for the treatment of osteoporosis in diffuse connective tissue diseases in children: a prospective multicenter study. Arthritis Rheum. 2000 Sep;43(9):1960-6. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-J. PMID 11014345
- [Background] Brumsen C, Hamdy NA, Papapoulos SE. Long-term effects of bisphosphonates on the growing skeleton. Studies of young patients with severe osteoporosis. Medicine (Baltimore). 1997 Jul;76(4):266-83. doi: 10.1097/00005792-199707000-00005. PMID 9279333
- [Background] Glorieux FH, Bishop NJ, Plotkin H, Chabot G, Lanoue G, Travers R. Cyclic administration of pamidronate in children with severe osteogenesis imperfecta. N Engl J Med. 1998 Oct 1;339(14):947-52. doi: 10.1056/NEJM199810013391402. PMID 9753709
- [Derived] Bianchi ML, Colombo C, Assael BM, Dubini A, Lombardo M, Quattrucci S, Bella S, Collura M, Messore B, Raia V, Poli F, Bini R, Albanese CV, De Rose V, Costantini D, Romano G, Pustorino E, Magazzu G, Bertasi S, Lucidi V, Traverso G, Coruzzo A, Grzejdziak AD. Treatment of low bone density in young people with cystic fibrosis: a multicentre, prospective, open-label observational study of calcium and calcifediol followed by a randomised placebo-controlled trial of alendronate. Lancet Respir Med. 2013 Jul;1(5):377-85. doi: 10.1016/S2213-2600(13)70064-X. Epub 2013 Jun 2. PMID 24429202
- See also: Lab test information — http://www.lios.it/research/telethon/Bianchi_CF-protocol-2000-labtests.pdf